CLINICAL TRIAL: NCT01629550
Title: Prospective Randomized Controlled Multicenter Trial of 4 Antiseptic Strategies for Prevention of Catheter Infection in Intensive Care Unit for Adults Patients
Acronym: CLEAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CLEAN
Record Dates: First submitted 2012-06-20; First posted 2012-06-27 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2014-03

CONDITIONS: Preventing Catheter Related Infection

ARMS (4):
- PVI paint (Active Comparator): 5% alcoholic povidone iodine paint
  Interventions: Procedure: skin disinfection prior catheter insertion
- PVI scrub and paint (Active Comparator): detersion with 4% povidone iodine scrub followed by 5% alcoholic povidone iodine paint
  Interventions: Procedure: skin disinfection prior catheter insertion
- Chlorhexidine paint (Active Comparator): 2% alcoholic chlorhexidine paint
  Interventions: Procedure: skin disinfection prior catheter insertion
- chlorhexidine scrub and paint (Active Comparator): Detersion with 4% chlorhexidine scrub followed 2% alcoholic chlorhexidine paint
  Interventions: Procedure: skin disinfection prior catheter insertion

INTERVENTIONS:
Procedure: skin disinfection prior catheter insertion

SUMMARY:
Catheter related infection is the third cause of nosocomial infection in ICUs. Most of them are avoidable and can be prevent by improving aseptic practices during catheter insertion and maintenance. Indeed, the main route of catheter contamination for short-term catheters is the insertion site. Consequently, the quality of skin disinfection is the most effective preventive measure to reduce the incidence of these infections.

This aim of the present study is to compare four strategies of skin disinfection to determine whether a 2% alcoholic solution of chlorhexidine acts better than 5% alcoholic povidone iodine in reducing catheter infection and to assess whether a detersion phase prior to disinfection reduces catheter colonization as compared with no detersion.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 year-old
* Expected duration of ICU stay ≥ 48 hours
* Patient requiring the insertion of at least one arterial catheter and/or central venous catheter and/or catheter for hemodialysis.

Exclusion Criteria:

* Patient with history of allergy to any of the antiseptic agent studied
* Expected survival < 48 hours
* Catheter inserted outside the ICU or in emergency without respect of preventive measures.
* Use of antimicrobial impregnated catheters or antiseptic impregnated dressings.
* Pregnant woman or breast-feeding mother

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400
Dates: Start 2012-10

PRIMARY OUTCOMES:
Major catheter related infection

SECONDARY OUTCOMES:
Catheter colonization
Catheter related bacteremia
Colonization insertion site
Prolongation hospitalization due to catheter infection
Mortality due to catheter infection
Skin allergy and anaphylactic shock
Costs

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Angers University Hospital, Angers
  - Estain University Hospital, Clermont-Ferrand
  - Bichat-Claude Bernard Hospital, Paris
  - Lyon University Hospital, Pierre-Bénite
  - Poitiers University Hospital, Poitiers

REFERENCES:
- [Derived] Iachkine J, Buetti N, de Grooth HJ, Briant AR, Mimoz O, Megarbane B, Mira JP, Valette X, Daubin C, du Cheyron D, Mermel LA, Timsit JF, Parienti JJ. Development and validation of a multivariable model predicting the required catheter dwell time among mechanically ventilated critically ill patients in three randomized trials. Ann Intensive Care. 2023 Jan 16;13(1):5. doi: 10.1186/s13613-023-01099-9. PMID 36645531
- [Derived] Iachkine J, Buetti N, de Grooth HJ, Briant AR, Mimoz O, Megarbane B, Mira JP, Ruckly S, Souweine B, du Cheyron D, Mermel LA, Timsit JF, Parienti JJ. Development and validation of a multivariable prediction model of central venous catheter-tip colonization in a cohort of five randomized trials. Crit Care. 2022 Jul 7;26(1):205. doi: 10.1186/s13054-022-04078-x. PMID 35799302
- [Derived] Buetti N, Ruckly S, Lucet JC, Bouadma L, Schwebel C, Mimoz O, Timsit JF. Ultrasound guidance and risk for intravascular catheter-related infections among peripheral arterial catheters: a post-hoc analysis of two large randomized-controlled trials. Ann Intensive Care. 2020 Jul 8;10(1):89. doi: 10.1186/s13613-020-00705-4. PMID 32643100
- [Derived] Maunoury F, Farinetto C, Ruckly S, Guenezan J, Lucet JC, Lepape A, Pascal J, Souweine B, Mimoz O, Timsit JF. Cost-effectiveness analysis of chlorhexidine-alcohol versus povidone iodine-alcohol solution in the prevention of intravascular-catheter-related bloodstream infections in France. PLoS One. 2018 May 25;13(5):e0197747. doi: 10.1371/journal.pone.0197747. eCollection 2018. PMID 29799871
- [Derived] Mimoz O, Lucet JC, Kerforne T, Pascal J, Souweine B, Goudet V, Mercat A, Bouadma L, Lasocki S, Alfandari S, Friggeri A, Wallet F, Allou N, Ruckly S, Balayn D, Lepape A, Timsit JF; CLEAN trial investigators. Skin antisepsis with chlorhexidine-alcohol versus povidone iodine-alcohol, with and without skin scrubbing, for prevention of intravascular-catheter-related infection (CLEAN): an open-label, multicentre, randomised, controlled, two-by-two factorial trial. Lancet. 2015 Nov 21;386(10008):2069-2077. doi: 10.1016/S0140-6736(15)00244-5. Epub 2015 Sep 18. PMID 26388532
- [Derived] Goudet V, Timsit JF, Lucet JC, Lepape A, Balayn D, Seguin S, Mimoz O. Comparison of four skin preparation strategies to prevent catheter-related infection in intensive care unit (CLEAN trial): a study protocol for a randomized controlled trial. Trials. 2013 Apr 27;14:114. doi: 10.1186/1745-6215-14-114. PMID 23782845